CLINICAL TRIAL: NCT02310893
Title: Effectiveness of Peer Navigation and Contingency Management on Retention in HIV Care
Acronym: CHAMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01MH103076-01A1 (NIH)
Record Dates: First submitted 2014-07-18; First posted 2014-12-08 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Contingency Management only (Active Comparator): Participants assigned to this arm will receive payments for attending regular HIV medical appointments at the clinic and filling prescribed HIV medications at the pharmacy
  Interventions: Behavioral: Contingency Management
- Peer Navigation only (Active Comparator): Participants in this arm will be assigned a peer navigator to assist them in accessing and remaining in HIV care
  Interventions: Behavioral: Peer Navigation
- Combined Contingency Management and Peer Navigation (Experimental): Participants in this arm will be assigned a peer navigator to assist them in accessing and remaining in HIV care and will be eligible to receive incentives for attending HIV care visits/refilling prescriptions.
  Interventions: Behavioral: Combined Contingency Management and Peer Navigation
- Usual care (No Intervention): Participants in this arm will receive the care that they would usually get in their clinic in the absence of this study.

INTERVENTIONS:
Behavioral: Combined Contingency Management and Peer Navigation
  Arms: Combined Contingency Management and Peer Navigation
Behavioral: Contingency Management
  Arms: Contingency Management only
Behavioral: Peer Navigation
  Arms: Peer Navigation only

SUMMARY:
Consistent treatment with anti-retroviral therapy (ART) suppresses viral load (VL), prolonging life and improving quality of life for HIV+ persons. Suppressing VL benefits communities by reducing transmission to others. Mere availability of ART and care, however, is insufficient; the benefits of ART depend upon HIV+ persons' continuous visits to the health care provider, regular monitoring and regular delivery of medications, - known as retention in HIV care. In spite of national efforts, up to a quarter of HIV+ persons, especially low-income minorities are out of care. Innovative interventions are therefore urgently needed to maximize engagement and retention in HIV care, self-reported adherence, as well as HIV-1 RNA viral load suppression. In pursuit of these aims, the proposed study will assess outcomes of the following interventions in comparison to usual care: 1) contingency management (CM) only; 2) peer navigation (PN) only; and 3) a combined approach that integrates both CM and PN (CA) which the investigators hypothesize to be most effective in improving HIV clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed HIV+
2. Age 18 years or older
3. English or Spanish speaking
4. Residence in Los Angeles County
5. prescribed ART in prior 24 months
6. < 3 visits in prior 12 months or have detectable viral load, as identified in the Ryan White CaseWatch database

Exclusion Criteria:

Not meeting any of the criteria identified above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2016-01; Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Change in retention-in-care behaviors over 12 months | Basline, follow-ups at month 2, 6, 12
  Using a 2x2 factorial design, to examine the effect of the three interventions -- peer navigation, contingency management, combined approach and usual care -- and evaluate how well they improve retention in HIV care
Change in HIV RNA viral load suppression and medication adherence over 12 months | Basline, follow-ups at month 2, and 12
  Using the same design, to examine the effects of the PN, CM and, CA interventions on HIV RNA viral load suppression and self-reported adherence

SECONDARY OUTCOMES:
Cost effectiveness | 5 years
  A secondary aim is to examine the cost-offset and potential cost-effectiveness of each intervention compared with usual care

CONTACTS AND LOCATIONS:
Overall Officials: William Cunningham, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (6):
- United States (6):
  - Center for Health Justice, Los Angeles, California
  - Los Angeles Sheriff's Department, Los Angeles, California
  - AltaMed Health Services Corporation, Los Angeles, California
  - Oasis Clinic, Los Angeles, California
  - Olive View Medical Center, Sylmar, California
  - Northeast Valley Health Corporation, Van Nuys, California